CLINICAL TRIAL: NCT04636944
Title: Learning From Heart Failure Nurses and Patients: Exploring Their Perspectives in the Management of Depression and Anxiety in Primary Care Settings
Brief Title: Management of Depression and Anxiety in HF
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID: 268951
Record Dates: First submitted 2020-10-28; First posted 2020-11-19 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure; Depression; Anxiety
MeSH Terms: conditions — Heart Failure; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: web-based COMPASS intervention — COMPASS is a web-based intervention (online CBT program) that was developed for managing illness-related anxiety and depression in patients with long-term conditions (LTC) (https://compass-ltc.org/). COMPASS is tailored to gain an understanding of the difficulties that LTC patients experience and provide information and tools on how to manage these. This qualitative study will explore participants' perspectives on using COMPASS for managing depression and anxiety in heart failure.

SUMMARY:
Heart failure (HF) is a complex clinical syndrome characterized by inability of the heart to pump an adequate amount of blood. Heart failure affects patients' ability to carry out even simple activities of daily living and therefore has negative psychological impact. Many studies reported that depression is prevalent among HF patients and it is being associated with high morbidity, mortality and costs. The European Society of Cardiology guidelines stresses the importance of routine depression screening with a validated questionnaire and initiating treatment for depression for all depressed HF patients and their access to psychological treatment.

The community heart failure nurses provide the integrated heart failure service in the local area of Southwark and Lambeth in South London. The aim of the integrated heart failure team in the community is to provide the HF treatment effectively, help patients understand and manage their symptoms and support with lifestyle changes. Even though, the community HF nurses have extensive role in managing HF patients in the community, their role in assessing anxiety and depression; and providing psychological treatment needs to be further explored.

Therefore, there is a need to assess the process by which community HF nurses assess and manage anxiety and depression. This current study builds on our recent systematic review which illustrated how cognitive behaviour therapy is effective at improving depressive symptoms in HF, but more studies are needed to build on these findings. The findings from this review will be used to examine the perspectives on assessing, managing and treating depression and anxiety in HF patients.

In this current study, an online focus group with community heart failure nurses and qualitative telephone/online interviews with community-based HF patients will be undertaken to explore their views and experiences in managing depression and anxiety; and to assess whether COMPASS a web-based intervention would be useful. Also, this study will explore the impact of COVID-19 on the psychological wellbeing of community-based HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for Community-based HF patients:

  1. Community-based HF patients with clinically established HF diagnosis (confirmed HF diagnosis) in Lambeth and Southwark Boroughs who have mild to moderate symptoms of depression with/without anxiety confirmed by PHQ-9 (5-14) and GAD-7;
  2. Patients with NYHA class I-III;
  3. Capacity to provide informed consent; and
  4. Proficiency in English language so can fully respond to verbal and written material.

Inclusion criteria for Community HF nurses:

1. All community-based HF-nurses employed in Lambeth and Southwark Boroughs who are registered with Nursing Midwifery Council (NMC) will be invited to participate in the study;
2. Capacity to provide informed consent;
3. Community HF-nurses who are actively providing care to community-based HF patients; and
4. have access to internet connected computer or device and technology for Microsoft (MS) Teams.

Exclusion Criteria:

* Exclusion criteria for community-based HF patients:

  1. Community-based HF patients under 18 years of age;
  2. Participants who are deemed not to have the capacity to consent;
  3. Patients with cognitive impairment or dementia confirmed by medical records; and
  4. Community-based HF patients with NYHA class IV.
  5. Patients with severe depression and/or having suicidal ideation.

Exclusion criteria for Community HF nurses:

1. Nurses working with inpatients or in the OPD departments; and
2. Nurses who are not employed as community HF nurses.
3. Any community HF nurse who do not have access to internet or online technology.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Guys and St. Thomas's community-based HF services in Lambeth and Southwark Boroughs.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Explore community heart failure nurses' perception of assessing, managing and treating depression and anxiety in HF and the use of web-based interventions. | This will take place before the introduction of COMPASS web-based intervention.
  will explore nurses' perception regarding the assessment and management of depression and anxiety in heart failure by undertaking an online focus group with community heart failure nurses.
Explore community heart failure patients' perception of assessing, managing and treating depression and anxiety in HF and the use of web-based interventions. | This will take place before the introduction of COMPASS web-based intervention.
  will explore patients' perception regarding the assessment and management of depression and anxiety in heart failure. This will be done by undertaking online\telephone interviews with community-based heart failure patients.
Explore nurses' perception of using web-based COMPASS intervention for depression and anxiety management in HF | This will take place 30 minutes after the introduction and demonstration of COMPASS web-based intervention.
  will explore nurses' perception regarding the use of web-based COMPASS intervention for the management of depression and anxiety in heart failure in an online focus group.
Explore patients' perception of using web-based COMPASS intervention for depression and anxiety management in HF | This will take place 30 minutes after the introduction and demonstration of COMPASS web-based intervention.
  will explore patients' perception regarding the use of web-based COMPASS intervention for the management of depression and anxiety in heart failure. This will be done by conducting online\telephone interviews with community-based heart failure patients.

SECONDARY OUTCOMES:
Explore with community HF nurses the impact of COVID-19 pandemic on HF patients' depression and anxiety level and changes to management processes. | This will take place before the introduction of COMPASS web-based intervention.
  will discuss with community HF nurses the impact of COVID-19 on the psychological wellbeing of community-based HF patients and how it changed their access to psychological intervention. This will form part of the online focus group.
Explore with community HF patients the impact of COVID-19 pandemic on HF patients' depression and anxiety level and changes to management processes. | This will take place before the introduction of COMPASS web-based intervention.
  will explore with community HF patients the impact of COVID-19 on the psychological wellbeing of community-based HF patients and how it changed their access to psychological intervention. This will form part of the online/telephone interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Silapiya Smith, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Catherine Evans, Study Director — Cicely Saunders Institute of Palliative Care, Rehabilitation and Policy, Faculty of Nursing, Midwifery and Palliative Care, King's College London,
Locations (1):
- Community Heart Failure Team: Elmcourt Health Centre, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT04636944/Prot_000.pdf